CLINICAL TRIAL: NCT03081338
Title: A Programme for Amyotrophic Lateral Sclerosis Care in Europe
Acronym: ALS-CarE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH18567
Record Dates: First submitted 2015-11-16; First posted 2017-03-16 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis); MND (Motor Neurone DIsease)
Keywords: ALS, MND, Care, Patient journey
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: A mix of incident and prevalent patient cases will be included in order to capture patients at different stages of the disease trajectory.

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) or else known as Motor Neurone Disease (MND) is a rapidly progressive fatal neurological disease that strikes in the prime of life, and for which there is no treatment. The principal aim of management is to maintain quality of life and reduce the symptoms of the disease. This requires a multidisciplinary approach using best practice for symptom alleviation, including innovation approaches towards maximising quality of life. The purpose of this study is to use existing information drawn from partner countries into a system of care that is available to people with amyotrophic lateral sclerosis at the correct time, in the correct format and in a cost effective manner. This will be achieved by collecting details of patient and carer experiences across all stages of from diagnosis to end of life, including decision making in the terminal stages of the disease. A health economic analysis will help to identify the overall costs of disease management, provide models of increased efficiency that preserve and maximize quality of life, and begin to develop novel health economic measurement tools for terminal neurological illness. The completed project will provide a user-friendly best practice programme for amyotrophic lateral sclerosis that can be modified for management of other related degenerative diseases of the nervous system.

DETAILED DESCRIPTION:
This is a prospective multi-centre observational research project that will be carried out by 8 European partners in 9 sites: 1 in Ireland (Dublin), 1 in the Netherlands (Utrecht), 2 in the United Kingdom (UK) (Sheffield and London), 2 in Italy (Turin and Milan), 2 in Germany (Berlin and Munich), and 1 in Belgium (Leuven). In terms of data collection, the study consists of 3 substudies and will be organised in 6 interlinked work packages spanning clinical, epidemiological and health services research.

All partners will contribute in participant recruitment and collect comparable data, which will be used for fulfilling the deliverables of each work package. Central co-ordination of research activities in the 2 UK sites will be undertaken in Sheffield. This protocol concerns research activities in relation to the ALS-CarE project involving the 2 UK-based participating sites.

Following ethical and research governance approvals, ALS-CarE officially started on 1st April 2014 and will run for 3 years. Participant recruitment will commence following ethical and research governance approval and will occur for the first 4 months at the Sheffield and King's College MND Care Centres. The follow-up period of each participant will take 12 months depending on the rate of progression of the illness. Finally, a period of 11 months at the end of the project will enable analysis of data, dissemination of findings and report writing.

SCIENTIFIC SUMMARY

Background:

Amyotrophic Lateral Sclerosis (ALS) or else known as Motor Neurone Disease (MND) is a progressive neurodegenerative disease that strikes in the prime of life. There are currently no effective disease modifying therapies for ALS and death usually occurs within 3 years of symptom onset. Management is palliative and is aimed at maximising quality of life and minimising the burden of disease. The complexity and rapidly progressive nature of ALS requires a responsive multidisciplinary care system that that is built on reliable disease staging and evidence based symptom management.

Aim:

To incorporate detailed clinical information drawn from population based sources into a responsive care programme.

Plan of investigation:

A standardised staging system will be validated, and quality of life and patient experiences will be measured and management optimised across disease stages from diagnosis to end of life. Health economic analysis will identify key differences in resource utilisation and will be useful for pharmaco-economic analyses of new therapeutics.

Potential impact:

The completed project will provide a user-friendly best practice framework for ALS that can be modified for management of other neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of definite, probable, laboratory supported or possible ALS according to the El Escorial criteria.

Exclusion Criteria:

* Patient cognitive impairment to the extent that they cannot complete an informed consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A mix of incident and prevalent cases will be included in order to capture patients at different stages of the disease trajectory. The total study population will contain 600 patients (300 newly diagnosed and 300 prevalent).
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Calculation of quality-adjusted life years (QALYs) that are used to inform economic evaluations of health care interventions using the EuroQoL validated EQ-5D-5L questionnaire. | 4 years
  Two potential service changes will be identified through examination of the patient journey and through the review of discordance with existing best practice guidelines. Key areas of interest are likely to be focussed around the organisation and delivery of services for gastrostomy, non-invasive ventilation, management of cognitive and behavioural impairment, and the involvement of specialised palliative care teams. The precise methods used will be determined on consideration of the types of intervention and types of data available, but are likely to include case-matching and/or more sophisticated statistical methods such as logistic regression or propensity scoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Institute for Translational Neuroscience, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No